CLINICAL TRIAL: NCT04663750
Title: Vitrectomy, Subretinal Tissue Plasminogen Activator and Intravitreal Gas for Submacular Haemorrhage Secondary to Exudative Age-Related Macular Degeneration (TIGER): a Phase 3, Pan-European, Two-group, Observer-masked, Superiority, Randomised Controlled Surgical Trial.
Brief Title: Vitrectomy, Subretinal Tissue Plasminogen Activator (TPA) and Intravitreal Gas for Submacular Haemorrhage Secondary to Exudative (Wet) Age-related Macular Degeneration (TIGER).
Acronym: TIGER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); Fight for Sight (Funder) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS Project ID: 276366; 2020-004917-10 (EudraCT Number)
Record Dates: First submitted 2020-11-27; First posted 2020-12-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-07

CONDITIONS: Eye Diseases; Macular Degeneration, Wet; Sub-Macular Hemorrhage
Keywords: Macular Degeneration, Wet; Sub-Macular Hemorrhage
MeSH Terms: conditions — Eye Diseases; Wet Macular Degeneration | interventions — aflibercept; Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: Experimental arm: pars plana vitrectomy, sub retinal injection of recombinant tissue plasminogen activator (TPA), intravitreal sulfahexafluoride (SF6) gas tamponade and intravitreal aflibercept.
  Active comparator arm: intravitreal aflibercept.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Surgery with aflibercept (Experimental): Surgery with aflibercept at the end of surgery, with post-operative review day 1 and week 1 (day 7)
  Interventions: Procedure: Pars plana vitrectomy; Drug: Intravitreal 2 mg aflibercept (Eylea, Bayer) will be injected at baseline then monthly for two further doses, then 2-monthly until month 12; Drug: subretinal injection of recombinant TPA (Alteplase) up to a maximum of 25 micrograms in 0.2 mls; Drug: Intravitreal 20% sulfahexafluoride (SF6) gas tamponade
- Arm B - Aflibercept monotherapy (Active Comparator): Aflibercept monotherapy commencing at baseline.
  Interventions: Drug: Intravitreal 2 mg aflibercept (Eylea, Bayer) will be injected at baseline then monthly for two further doses, then 2-monthly until month 12

INTERVENTIONS:
Procedure: Pars plana vitrectomy — Pars plana vitrectomy
  Arms: Arm A - Surgery with aflibercept
Drug: Intravitreal 2 mg aflibercept (Eylea, Bayer) will be injected at baseline then monthly for two further doses, then 2-monthly until month 12 — Intravitreal 2 mg aflibercept (Eylea, Bayer) will be injected at baseline then monthly for two further doses, then 2-monthly until month 12.
  Other Names: Aflibercept (Eylea, Bayer)
Drug: subretinal injection of recombinant TPA (Alteplase) up to a maximum of 25 micrograms in 0.2 mls — Subretinal injection of recombinant TPA (Alteplase, Actilyse, Boehringer Ingelheim) up to a maximum of 25 micrograms in 0.2 mls.
  Other Names: Actilyse (Boehringer Ingelheim)
  Arms: Arm A - Surgery with aflibercept
Drug: Intravitreal 20% sulfahexafluoride (SF6) gas tamponade — Intravitreal 20% sulfahexafluoride (SF6) gas tamponade.
  Arms: Arm A - Surgery with aflibercept

SUMMARY:
The centre of the retina (macula) at the back of the eye contains cells that give us our central vision that we use for reading and recognising faces. These cells can be damaged by a disease called wet age-related macular degeneration (AMD), where new abnormal blood vessels grow through the macula and leak fluid. This can affect vision. In some cases, wet AMD can also cause a bleed under the macula, known as a submacular haemorrhage (SMH), which can lead to marked and persistent loss of vision in the eye.

The current standard treatment for wet AMD is to give injections containing 'anti-VEGF' drugs into the eye. Anti-VEGF drugs reduce the leakage of fluid so that the macula can become dry again and sight can improve.

Anti-VEGFs are also the current standard of care for SMH, mainly because there is no licensed treatment for the SMH itself (patients with SMH were excluded from most wet AMD studies).

The purpose of this study therefore is to compare two treatments:

1. Standard treatment for wet AMD (anti-VEGF injections).
2. Standard treatment above plus surgery. This study will find out if having surgery alongside anti-VEGF injections can improve vision further over the current standard treatment of anti-VEGF injections alone.

DETAILED DESCRIPTION:
SMH is a rare but devastating complication of wet AMD. Untreated, SMH typically leads to permanent and severe loss of vision, ranging from 6/30 (approximately 20% normal vision) to only being able to perceive light versus dark (no useful vision).

There are no large, published, randomised controlled trials (RCTs) evaluating treatments for SMH. Hence there is no widely-accepted treatment approach. Some patients are managed by observation, others with drugs (anti-VEGF) injected into the eye, others with eye surgery (vitrectomy, subretinal TPA, gas) and combinations thereof. From a regulatory perspective the standard treatment is with anti-VEGF injections alone, since these are licensed for the treatment of wet AMD (and there is no treatment licensed for SMH). This study will test the hypothesis that surgery with anti-VEGF injections for SMH due to wet AMD is superior to the current standard of treatment with anti-VEGF injections alone. The results will help guide future clinical practice to maximise the visual outcomes for patients with SMH. Most potential participants will present or be referred to the clinics of the investigators who provide routine care for wet AMD. Referrals may arise from research networks, family physicians, optometrists or ophthalmologists.

After confirming the diagnosis of SMH, informed consent will be obtained and potential participants will be asked to sign a consent form. Following this, baseline screening will occur, including a clinical examination and a series of vision tests to confirm eligibility to take part in the study.

Once successfully screened, each participant will be randomly allocated to one of the two study groups:

1. Standard current treatment with anti-VEGF injections: participants will be given their first injection into the study eye at the screening/baseline visit, or otherwise within a few days. Following this, each participant will receive another injection at month 1, another at month 2 and thereafter one injection every two months until the end of the study (month 12). Anaesthetic eye drops will be given to numb the eye before each injection.
2. Standard current treatment with anti-VEGF injections plus surgery: participants will be given their first injection into the study eye at the time of surgery and then all other injections as per the schedule above. During the surgery, the clear gel (vitreous) that fills the inside of the eye will be removed and a clot-busting drug (TPA) will be injected into the eye to help break up the blood clot. The inside of the eye will then be filled with gas to help push the dissolved clot away from the macula. Various options for anaesthetic will be discussed with each participant before surgery, including (i) local anaesthetic only, (ii) local anaesthetic with some sedation, to reduce any anxiety or (iii) general anaesthetic so the participant is asleep during the surgery. If the participant also has a cataract or is likely to develop one, the surgeon will discuss the option of having cataract surgery as part of the same operation.

After the surgery, participants will be asked to keep their heads forward, to enable the gas bubble to move the blood clot away from the macula. This should be done for 50 minutes out of every hour for the first five days. During the 10-minute breaks, participants will be encouraged to move around and be active. At night, participants will be asked to sleep on the side of the operated eye, i.e. with the operated eye lowest. The gas is expected to disappear from the eye around 4-8 weeks after surgery.

Participants who have had surgery will be instructed to return for follow up the day after surgery and also one week later. All participants will also have a clinical examination at 6 and 12 months that will include tests of their vision. They will also attend regularly for anti-VEGF injections: every month for the first three visits, then every two months until the study is completed at month 12.

ELIGIBILITY:
Inclusion Criteria:

General

1. Males or females aged at least 50 years

   Study eye
2. SMH, comprising sub-neuroretinal haemorrhage with or without sub-RPE haemorrhage, that occurs secondary to treatment naïve, or previously treated exudative AMD, including choroidal neovascularisation (CNV), idiopathic polypoidal choroidal vasculopathy (IPCV) and retinal angiomatous proliferation (RAP).
3. SMH involving the foveal centre that measures at least 1 disc diameter in greatest linear dimension.
4. Sub-neuroretinal haemorrhage at least 125 microns thick, measured at the foveal centre using spectral-domain optical coherence tomography (SD-OCT).
5. BCVA between counting fingers and an Early Treatment of Diabetic Retinopathy Study (ETDRS) letter score of 70, inclusive.

Exclusion Criteria:

General

1. Serious allergy to fluorescein or indocyanine green (ICG).
2. Hypersensitivity to alteplase, gentamicin, arginine, phosphoric acid, polysorbate 80 or aflibercept (Eylea).
3. Stroke, transient ischaemic attack or myocardial infarction within 6 months.
4. Participation in another interventional study within 12 weeks of enrolment or planned to occur during this study.
5. Women who are breast feeding, pregnant, or planning to become pregnant during the clinical trial. Any sexually active women of childbearing potential must agree continued abstinence from heterosexual intercourse or to use highly effective methods of birth control for the duration up to 12 weeks after administration of IMP or the last administration of aflibercept on the trial. Men must also agree to use a condom if their partner is of child bearing potential, even if they have had a successful vasectomy. Females of childbearing potential are females who have experienced menarche and are not surgically sterilised (e.g. hysterectomy or bilateral salpingectomy) or post-menopausal (defined as at least 1 year since last regular menstrual period). Highly effective methods of birth control are those with a failure rate of < 1% per year when employed consistently and correctly, eg. combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation via oral, intravaginal, and transdermal routes; progestogen-only hormonal contraception associated with inhibition of ovulation via oral, injectable, implantable, intrauterine device (IUD), or intrauterine hormone-releasing system ( IUS); or vasectomised partner.
6. International Normalised Ratio (INR) greater than 3.5, unless it is anticipated that the INR can be brought below this level prior to vitrectomy, balancing the systemic risks with those of intraocular haemorrhage*.
7. Unwilling, unable, or unlikely to return for scheduled follow-up for the duration of the trial.
8. Any other condition which, in the opinion of the investigator, would prevent the participant from granting informed consent or complying with the protocol, such as dementia, mental illness, or serious systemic medical disease.

   Study eye
9. SMH that is known or estimated to have been present for longer than 15 days, as evidenced by history, pre-trial clinical documentation, or fundus appearance.
10. SMH due to eye disease other than exudative AMD.
11. Current active proliferative diabetic retinopathy.
12. Current intraocular inflammation.
13. Current ocular or periocular infection other than blepharitis.
14. Current or known former high myopia (>6 dioptres).
15. Aphakia.
16. Other current or pre-existing ocular conditions that, in the opinion of the Investigator, will preclude any improvement in BCVA following resolution of SMH, such as severe central macular atrophy or fibrosis, dense amblyopia, macular hole involving the fovea, or very poor BCVA prior to presentation with SMH (counting fingers or worse).
17. Inadequate pupillary dilation or significant media opacities, which will prevent adequate clinical evaluation of the posterior segment or fundus imaging.
18. Intraocular surgery within 12 weeks of enrolment except for uncomplicated cataract surgery, which is permitted within 8 weeks of enrolment.

    * Applies only to participants receiving warfarin.

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
assessment of Early Treat of Diabetic Retinopathy Study (ETDRS) letters of best-corrected visual acuity (BCVA) in the study eye. | 12 months
  The primary outcome is the proportion of participants with a BCVA gain ≥10 ETDRS letters in the study eye at the 12 month visit.

SECONDARY OUTCOMES:
Assessment of Early Treatment Diabetic Retinopathy Study (ETDRS) letter improvement in Best-Corrected Visual Acuity (BCVA) in the study eye | 6 months
  Change in ETDRS letters in BCVA in the study eye at the month 6 visit.
Mean ETDRS BCVA | 6 and 12 months
Radner maximum reading speed | 6 and 12 months
Area of scotoma size using Humphrey Field Analyser 10-2 or equivalent | 6 and 12 month
National Eye Institute 25-item visual function questionnaire (NEI VFQ-25). composite score. | 6 and 12 months.
EQ-5D-5L with vision bolt-on score. | 6 and 12 months.
Presence/absence of subfoveal fibrosis and/or atrophy and area of fibrosis/atrophy using multimodal reading centre image analysis. | 12 months.
  Presence or absence of subfoveal fibrosis and/or atrophy and area of fovea-involving fibrosis/atrophy assessed using multimodal imaging by an independent reading centre, combining spectral domain optical coherence tomography (SD-OCT), fundus autofluorescence (FAF) and stereo fundus photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Jackson, PhD, FRCOphth, Principal Investigator — Kings College London & Kings College Hospital
Locations (36):
- Germany (7):
  - University of Bonn, Bonn
  - University Medical Center Hamburg Eppendorf, Hamburg
  - Ludwig Maximilians-University München, München
  - Augenzentrum am St. Franziskus-Hospital Münster, Münster
  - Knappschaft Kliniken Saar GmbH, Sulzbach, Sulzbach
  - Ulm University Hospital, Ulm
  - University hospital of Würzburg, Würzburg
- The Institute of Eye Surgery, Waterford, Ireland
- Ophthalmology Clinic Jasne Błonia, Lodz, Poland
- University Hospital Bern, Bern, Switzerland
- United Kingdom (26):
  - Mid and South Essex NHS Foundation Trust, Chelmsford, Essex
  - Kent & Canterbury Hospital (East Kent University), Canterbury, Kent
  - King's College Hospital NHS Foundation Trust, London, London
  - The Princess Alexandra Eye Pavilion, Edinburgh, Scotlan
  - Sunderland Eye Infimary, Sunderland, Tyne and Wear
  - Hull Royal Infirmary, Hull, Yorkshire
  - Belfast Health and Social Care Trust, Belfast
  - University Hospitals Sussex NHS Trust, Brighton
  - Bristol Eye Hospital, Bristol
  - Royal Devon and Exeter Hospital, Exeter
  - Gartnavel General Hospital, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - Barts Health NHST trust - Whipps Cross University Hospital, London
  - Moorfields Eye Hospital, London
  - Imperial College Healthcare NHS Foundation Trust (The Western Eye Hospital), London
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - Manchester Royal Eye Hospital, Manchester
  - James Cook University Hospital, (South Tees NHSFT), Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHST, Plymouth
  - University Hospital Southampton NHS foundation Trust, Southampton
  - Torbay and South Devon NHS, Torquay
  - New Cross Hosp, Royal Wolverhampton NHST, Wolverhampton

REFERENCES:
- [Derived] Lee CN, Desai R, Ramazzotto L, Wafa H, Wang Y, Bunce C, Doungsong K, Ezeofor V, Edwards RT, Lois N, Steel DH, Peto T, Hillenkamp J, van Meurs JC, Reeves BC, Jackson TL. Vitrectomy, subretinal Tissue plasminogen activator and Intravitreal Gas for submacular haemorrhage secondary to Exudative Age-Related macular degeneration (TIGER): update to study protocol and addition of a statistical analysis plan and health economic analysis plan for a randomised controlled surgical trial. Trials. 2025 Apr 14;26(1):131. doi: 10.1186/s13063-025-08727-8. PMID 40229856
- [Derived] Jackson TL, Bunce C, Desai R, Hillenkamp J, Lee CN, Lois N, Peto T, Reeves BC, Steel DH, Edwards RT, van Meurs JC, Wafa H, Wang Y. Vitrectomy, subretinal Tissue plasminogen activator and Intravitreal Gas for submacular haemorrhage secondary to Exudative Age-Related macular degeneration (TIGER): study protocol for a phase 3, pan-European, two-group, non-commercial, active-control, observer-masked, superiority, randomised controlled surgical trial. Trials. 2022 Jan 31;23(1):99. doi: 10.1186/s13063-021-05966-3. PMID 35101110